CLINICAL TRIAL: NCT06754241
Title: Impact of Personalized Rehabilitation Guidance Based on WeChat Official Accounts Platform on Functional Recovery and Quality of Life of Patients with Knee Osteoarthritis
Brief Title: Impact of Personalized Rehabilitation Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yan Dong (Other)
Responsible Party: Sponsor-Investigator, Yan Dong, Principal Investigator, Fuyang Affiliated Hospital of Anhui Medical University
Organization: Fuyang Affiliated Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fuyang Affiliated Hospital 001
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Behavioral: conventional nursing care
- observation group (Experimental)
  Interventions: Behavioral: Intervention Care

INTERVENTIONS:
Behavioral: conventional nursing care — (1) Preoperative education: An appropriate walking aid was provided for the patient and instructions were given to guide correct use, while isometric muscle exercises were taught. (2) Postoperative care: Six hours after anesthesia recovery, the head of the patient's bed could be elevated as needed, and the patient was instructed to perform ankle pumps (dorsiflexion and plantarflexion of the ankle).(3) Postoperative exercise: One to two days after surgery, following the removal of the drainage tube, the patient was encouraged to continue with ankle pumps and isometric quadriceps contractions, as well as to begin straight-leg raises. (4) Postoperative Day 3: In strict accordance with medical advice and under the guidance of a physiotherapist, patients engaged in continuous passive motion therapy for the affected knee, along with manual knee joint massage. (5) Postoperative Days 5-7: the patient would try to stand with the assistance of a walker, gradually progressing to walking exercises
  Arms: control group
Behavioral: Intervention Care — (1) Intervention Day 1: (i) All patients in the observation group were provided with an introduction to the study and invited to join the WeChat group for the observation group. (2) Intervention Day 2: Exercise guidance for patients with KOA was shared via the WeChat group.(3) Intervention Day 3: Guidance for emotional regulation was sent to the patients with KOA via the WeChat group.(4) Intervention Week 1: A micro-lesson on KOA-related knowledge was delivered via the WeChat group to deepen patients' understanding. (5) Intervention Week 2: (i) Text instructions and related questions on common conservative treatments for KOA, including topical and oral painkillers, were shared, with correct answers provided the next day.(ii) A micro-lesson on exercise guidance for patients with KOA was uploaded to the WeChat group to reinforce patients' understanding.
  Arms: observation group

SUMMARY:
To investigate the impact of personalized rehabilitation guidance based on the WeChat Official Accounts Platform on the functional recovery and quality of life of patients with knee osteoarthritis (KOA).Ninety patients diagnosed with KOA undergoing joint replacement were included via convenient sampling.The patients were randomly divided into an observation group and a control group,with 45 patients in each group.The control group received traditional rehabilitation guidance,while the observation group received personalized rehabilitation guidance through the WeChat Official Accounts Platform in addition to the traditional guidance.Different care plans had varying effects on patients' scores on the 36-item Short Form Health Survey (SF-36),Visual Analog Scale (VAS),and Lysholm Knee Scoring Scale.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 to 80 years;
* conscious, without cognitive impairments, and able to complete reading independently or with assistance;
* able to operate a smartphone and use WeChat;
* willing to participate in this study and provide signed informed consent.

Exclusion Criteria:

* acute cerebrovascular disease with sequelae in the past 6 months;
* coexisting primary psychiatric disorders;
* unable to perform physical exercise due to physical disability in the lower limbs;
* postoperative complications, such as deep vein thrombosis or infection;
* participation in other interventional studies.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The 36-item Short Form Health Survey (SF-36) | at 1 week and 1 month post-discharge
  The SF-36 is a concise health survey divided into 8 subscales: physical function, role physical, bodily pain, global health, vitality, social function, role emotional, and mental health, where a higher score indicates a better health status.
Visual Analog Scale (VAS) | at 1 week and 1 month post-discharge
  The VAS was used to assess pain levels before and after treatment in the two groups. VAS scores are positively correlated with pain intensity, where 0 indicates no pain and 10 indicates the most severe pain. A score of ≤3 is defined as mild pain, 4-6 as moderate pain, and ≥7 as severe pain.
Lysholm Knee Scoring Scale | at 1 week and 1 month post-discharge
  The Lysholm Knee Scoring Scale was employed to evaluate knee function. This scale covers eight aspects, including limping, support, restraining, instability, pain, swelling, climbing stairs, and squatting. It is scored on a scale of 0 to 100. The total score is 100 points, with higher scores indicating fewer symptoms and higher levels of functioning. A score above 95 is considered excellent, 85-94 is good, 65-84 is fair, and less than 65 is poor.
The Newcastle Satisfaction with Nursing Scale (NSNS) | at 1 week and 1 month post-discharge
  The Newcastle Satisfaction with Nursing Scale (NSNS) was used to measure patient satisfaction with nursing care. This scale consists of 19 items, such as nurse competence, communication, emotional support, and safety management. Each item is rated on a scale of 1-5, with a total score ranging from 19 to 95 points. A score of ≥77 indicates very satisfied, 58-76 indicates satisfied, 39-57 indicates moderately satisfied, and ≤38 indicates dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuyang Hospital of Anhui Medical University, Fuyang, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Jiang S, Zhou M, Dong Y. WeChat-Based Personalized Rehabilitation: Enhancing Recovery and Quality of Life in Knee Osteoarthritis. Nurs Health Sci. 2025 Jun;27(2):e70149. doi: 10.1111/nhs.70149. PMID 40542658